CLINICAL TRIAL: NCT06225778
Title: The Effect of The 6 Week Online Exercise Program On Core Stability And Vertical Jump Performance In University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Collaborators: Yeditepe University (Other)
Responsible Party: Principal Investigator, Çağdaş IŞIKLAR, Physiotherapist, Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 01.03.2021
Record Dates: First submitted 2024-01-13; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2021-09

CONDITIONS: Exercise
Keywords: Core Stabilization, Vertical Jump, IPAQ-SF, MSPPA Exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Care Provider
Masking Description: Blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Control group
- Exercise Group (Experimental): 6-week online exercise group
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — 6-week online exercise group
  Arms: Exercise Group

SUMMARY:
The goal of this randomized controlled study is to examine the effect of the online exercise program on core stabilization and vertical jump performance and observe the relationship between physical activity levels and motivation. In addition, compare these parameters with the exercise group and control group. The main questions it aims to answer are:

Does a 6-week online exercise program at university have an effect on core stabilization and vertical jump? Does exercise have an effect on motivation and physical activity level?

DETAILED DESCRIPTION:
Background: The importance of physical activity and exercise is increasing day by day. The aim of this study is to examine the effect of the online exercise program on core stabilization and vertical jump performance and observe relationship with physical activity levels and motivation.

Methods: The study included 51 healthy volunteer students registered at Fenerbahçe University and actively continuing their education. Evaluations were made before the exercise program and at the end of the sixth week. All assessments and exercise program were conducted online. Two of Mcgill's trunk muscle endurance tests were preferred to evaluate core stability: Trunk extensor endurance test (TEET), bilateral side bridge endurance tests (SBET), and Prone Bridge Test (PBT) was preferred for flexor endurance. Vertical Jump (VJ) test was used to evaluate vertical jump height performance. The International Physical Activity Questionnaire-Short Form (IPAQ-SF) was used to determine the physical activity levels of individuals, and the Physical Activity Participation Motivation Scale (MSPPA) was used to measure their motivation to participate in physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Being an university student
* Having a good health
* Participant in ages between 18-27 years of age
* Participating to the study in a voluntary basis

Exclusion Criteria:

* Having had orthopedic surgery in the last 60 days
* Severe neurological or vestibular disease that would interfere with exercise
* Taking any medications that could affect balance

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Trunk extensor endurance test (TEET) | 0th and 6th Week
  Test time was recorded manually with a stopwatch. The longer stays in the same position, the better the test result.
Bilateral side bridge endurance tests (SBET) | 0th and 6th Week
  Test time was recorded manually with a stopwatch. The longer stays in the same position, the better the test result.
Prone Bridge Test (PBT) | 0th and 6th Week
  Test time was recorded manually with a stopwatch. The longer stays in the same position, the better the test result.
Vertical Jump Test | 0th and 6th Week
  Maximum jump height as an indicator of lower extremity muscle strength can provide important information about functional capacities and performances in most sports and people in preparation for sports

SECONDARY OUTCOMES:
Motivation Scale For Participation in Physical Activity | 0th and 6th Week
  The lowest score that can be obtained from the scale is 16 and the highest score is 80. Participants' high scores from the scale mean that their motivation to participate in physical activity is positive. In this context, the scores the participants receive from FAKMS are 1-16 for very low, 17-32 for low, 33-48 for medium, 49-64 for high, and 65-80 for very high physical activity. indicates that they have motivation to participate. 3rd, 9th, 13th, 14th, 15th, 16th of the scale. The items are inverse items.
International Physical Activity Questionnaire (IPAQ) | 0th and 6th Week
  Scoring a HIGH level of physical activity on the IPAQ means your physical activity levels equate to approximately one hour of activity per day or more at least a moderate intensity activity level.
  Scoring a MODERATE level of physical activity on the IPAQ means you are doing some activity more than likely equivalent to half an hour of at least moderate intensity physical activity on most days.
  Scoring a LOW level of physical activity on the IPAQ means that you are not meeting any of the criteria for either MODERATE of HIGH levels of physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Feryal Subaşı, Prof, Study Chair — Yeditepe University
Locations (1):
- Yeditepe University, Istanbul, Atasehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No